CLINICAL TRIAL: NCT03192683
Title: Patient and Parent Satisfaction With Sling Use After Pediatric Upper Extremity Fractures: A Randomized Controlled Trial
Brief Title: Modified "Providence" Pedi Cast-Sling vs.Cast and Sling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lifespan (Other)
Responsible Party: Principal Investigator, Aristides Cruz, Assistant Professor, Orthopaedic Surgery, Lifespan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 400316
Record Dates: First submitted 2017-06-18; First posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Fractures, Bone; Pediatric ALL
MeSH Terms: conditions — Fractures, Bone; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular sling (Active Comparator)
  Interventions: Device: Regular sling
- Cast-sling (Experimental)
  Interventions: Device: Providence Pedi Cast-Sling

INTERVENTIONS:
Device: Providence Pedi Cast-Sling — Custom made sling with readily available casting materials
  Arms: Cast-sling
Device: Regular sling
  Arms: Regular sling

SUMMARY:
Examining custom made sling vs. off the shelf sling for immobilization following pediatric upper extremity fractures.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 0-18 years old who were evaluated in the pediatric emergency department (ED) by the orthopaedic resident on call
* patients with an upper extremity fracture (wrist, forearm or elbow) that required placement of a long-arm cast.

Exclusion Criteria:

* open fractures
* fractures at multiple levels (e.g. wrist AND elbow fracture)
* fractures requiring immediate/urgent surgery
* patients requiring admission for any reason
* bivalved LAC's for any reason

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction scores | 1 week

IPD SHARING:
Plan to Share IPD: No